CLINICAL TRIAL: NCT02270502
Title: Ultrasound Assessment of Muscle to Quantify Frailty.
Brief Title: Effects of Frailty, Sarcopenia and Muscle Wasting on Outcomes of Patients in the Surgical Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Director of Research, Critical Care Division, Associate Professor of Anesthesia, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2014P000249
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Critical Illness; Sarcopenia; Muscle Wasting
Keywords: critically illness; intensive care unit; outcome; frailty
MeSH Terms: conditions — Critical Illness; Sarcopenia; Muscular Atrophy; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patients on the SICU: Adult patients on the surgical intensive care unit (SICU), within 72 hours of admission to the SICU and until SICU discharge. Ultrasound Philips CX50, Frailty Index questionnaire and muscle strength tests.
  Interventions: Device: Ultrasound Philips CX50; Other: Frailty Index Questionnaire; Other: Muscle strength tests

INTERVENTIONS:
Device: Ultrasound Philips CX50 — The Philips CX50 ultrasound system is used to measure muscle size of the patients. We will measure the area and diameter of the rectus femoris muscle via ultrasound.
Other: Frailty Index Questionnaire — Frailty Index Questionnaire is a clinical tool to assess frailty in patients. We will ask patients to answer the questionnaire, including clarification that the questionnaire assesses the patient's pre-admission condition. The presence of a frail characteristic will be scored as 1 point. Most variables will be dichotomized (e.g. 1 point when a frail characteristic will be present and 0 points when frail characteristic will be not present).The Frailty Index will be calculated as the total number of frail characteristics of the patient divided by the total number of variables (n=50).
Other: Muscle strength tests — MRC score is a clinical assessment of muscle power on abduction of the arm, flexion of the forearm, extension of the wrist, flexion of the leg, extension of the knee and dorsal flexion of the foot with the score of (0-5) on each measurement.

SUMMARY:
The primary aim of the study is to evaluate consequences of frailty in critically ill patients. We hypothesize that a higher frailty index (based on published questionnaires) predicts a longer surgical intensive care unit and hospital length of stay, less ventilator-free days and a higher likelihood of an adverse discharge disposition.

Our secondary aim is to identify muscle-size derived variables that can be used to predict frailty. We hypothesize that a low skeletal muscle mass measured by ultrasound can be used to quantify frailty, and to also predict the outcome of SICU patients, expressed as longer stay in the surgical intensive care unit and longer stay in the hospital, less ventilator-free days and a higher likelihood of an adverse discharge disposition.

Our third aim is to examine potential triggers of muscle wasting in critically ill patients. Muscle wasting will be assessed by repetitive ultrasound measurements of muscle mass. We hypothesize that a significant decrease in skeletal muscle mass predicts longer stay at the surgical intensive care unit and longer hospital length of stay, less ventilator-free days and adverse discharge disposition.

DETAILED DESCRIPTION:
Frailty is defined as status of decreased physiological reserve which leads to a higher vulnerability to stressors. It is associated with a higher risk of morbidity and mortality. Within the geriatric population, frailty is common and a known predictor of adverse outcomes. The usefulness of a frailty assessment as an outcome measure in critically ill patients of all ages needs to be evaluated. This study evaluates whether frailty has an effect on outcome of critically ill patients.

Muscle weakness predicts outcome of ICU patients but is hard to determine in the ICU since the measurement is volition dependent. Muscle mass correlates with muscle weakness and can be assessed objectively. This study evaluates the consequences of reduced muscle mass or sarcopenia on the outcome of critically ill patients.

In addition, muscle wasting in the ICU may predict persistent functional disability. This study aims to examine muscle wasting of critically ill patients on the surgical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the SICU (within 72 hours of admission)
* Age over 18 years
* Stay on the SICU for at least 24 hours

Exclusion Criteria:

* Ongoing discussions about goals of care
* Motor component of Glasgow Coma Scale <5
* Unstable fractures
* Preexisting paralysis
* Pregnancy
* Absence of both lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the surgical intensive care unit (SICU)
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Surgical intensive care unit length of stay | Patients will be followed until SICU discharge, an expected 2 days to 2 weeks.
  Time from study inclusion to SICU discharge, an expected time of 2 days to 2 weeks.

SECONDARY OUTCOMES:
Hospital length of stay | Patients will be followed until hospital discharge, an expected 4 days to 4 weeks
  Time from study inclusion to hospital discharge, an expected time of 4 days to 4 weeks
Discharge Disposition | Patient will be followed until hospital discharge, an expected 4 days to 4 weeks
  Discharge disposition of the patient expressed as home, rehabilitation, nursing facility or in-hospital mortality.
Ventilator-free days | Patients will be followed until SICU discharge, an expected 2 days to 2 weeks.
  Days spent on the SICU that patient is not receiving mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mueller N, Murthy S, Tainter CR, Lee J, Riddell K, Fintelmann FJ, Grabitz SD, Timm FP, Levi B, Kurth T, Eikermann M. Can Sarcopenia Quantified by Ultrasound of the Rectus Femoris Muscle Predict Adverse Outcome of Surgical Intensive Care Unit Patients as well as Frailty? A Prospective, Observational Cohort Study. Ann Surg. 2016 Dec;264(6):1116-1124. doi: 10.1097/SLA.0000000000001546. PMID 26655919